CLINICAL TRIAL: NCT01527994
Title: Clinical Laboratory Evaluations of Aprepitant for the Treatment of Opioid Dependence: Inpatient Test
Brief Title: Aprepitant Effects in Intravenous Heroin Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-0457; 5R01DA027151-02 (NIH)
Record Dates: First submitted 2012-01-09; First posted 2012-02-07 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Opioid Dependence
Keywords: Aprepitant; Intravenous heroin dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant 125 mg (Experimental): Day Number Dose Procedure Day 0 Aprepitant 125mg Admitting Medication Treatment Day 1 Aprepitant 125mg Saline-Saline Day 2 Aprepitant 125mg Morphine-Morphine Day 3 Aprepitant 125mg Saline-Morphine Day 4 Aprepitant 125mg Naloxone-Morphine and Discharge
  Interventions: Drug: Aprepitant
- Placebo (Placebo Comparator): Day Number Dose Procedure Day 0 placebo Admitting Medication Treatment Day 1 placebo Saline-Saline Day 2 placebo Morphine-Morphine Day 3 placebo Saline-Morphine Day 4 placebo Naloxone-Morphine and Discharge
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Aprepitant — Aprepitant 125 mg oral tablets
  Other Names: Brand name: Emend
  Arms: Aprepitant 125 mg
Drug: Placebo pill — Placebo oral pill- inactive compound
  Arms: Placebo

SUMMARY:
Current treatments for opioid addiction would benefit by the addition of a non-opioid based treatment medication. Recent behavioral studies have shown that the neurokinin-1 (NK1) receptor is involved in opioid reward and withdrawal. This study proposes to study a potential non-opioid treatment, the clinically available, FDA approved, NK1 antagonist aprepitant, in opioid addicted patients. Based on the unique behavioral and pharmacological characteristics of opioid addiction, and what is known of the currently employed treatments, the investigators propose that the therapeutic mechanism of any potential opioid addiction treatment medication must include the ability to reduce opioid withdrawal. This is of particular importance during treatment initiation (eg. detoxification). In addition, for long-term treatment and relapse prevention, it is important to manage drug craving and inhibit the rewarding effects of opioids if patients do experience a slip. Therefore, the investigators propose to study aprepitant using human models of opioid withdrawal, craving and acute opioid reward and reinforcement. The investigators will also include a neuro-economics choice procedure paradigm.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ranging in age from 18-55 years who are currently opioid dependent based on meeting DSM-IV criteria for dependence on heroin and who are either treatment or non-treatment seeking individuals.
2. Use of intravenous heroin daily for a minimum of 45 days prior to study entry.
3. Urine sample (+) for opioids and prior experience with i.v. drug injection.
4. Female subjects who are not of childbearing potential, (i.e. post-hysterectomy, or two years post-menopausal) or who are of childbearing potential but will either abstain from heterosexual intercourse and/or practice a medically accepted form of contraception for the study duration.
5. Subjects who have experienced significant opioid withdrawal and are familiar with its effects.
6. Subjects who are willing to follow the protocol requirements, including methadone and study medication schedules, as evidenced by written informed consent and an ability to read, understand, and complete the study questionnaires.

Exclusion Criteria:

1. Subjects with any significant current axis-1 psychiatric problems, other than those related to drug abuse and opioid dependence, based on a structured psychiatric interview, SCID or MINI, during the screening process.
2. Subjects undergoing active treatment for any illness other than chronic stable medical conditions (Patients with HIV and/or taking anti-viral HIV medication without a manifestation of AIDS symptoms are allowed).
3. Subjects with clinically significant abnormal findings as determined by medical history, physical examination, vital signs (blood pressure, heart rate, and respiration rate), 02 saturation measure,12-lead ECG, clinical laboratory tests (CBC, chemistry panel), urine drug screen, alcohol breath test, and urine pregnancy test (for females of childbearing potential only).
4. Subjects who have any acute organ dysfunction or serious unstable disease states including symptomatic heart, renal or liver disease, COPD, sleep apnea, or encephalitis.
5. Subjects with 02 saturation below 90% at screening.
6. Subjects taking any concomitant medications (prescription and over-the-counter therapy) including psychotropic medications for the treatment of current major depression, schizophrenia, or mood disorders, as well as medications contraindicated for use with morphine, naltrexone, aprepitant, or methadone.
7. Subjects who have received any investigational drug or treatment within the thirty (30) days preceding administration of study medication.
8. Females who are nursing, pregnant (as confirmed by a positive urine pregnancy test), or at risk of becoming pregnant.
9. Subjects allergic or intolerant to morphine, methadone, naloxone, or aprepitant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Opioid Withdrawal | 30 minutes pre-medication, 150 minutes post medication, 15 minutes post-challenge drug administration, 1 hour post- challenge drug administration, 2 hours post challenge drug administration and 3.5 hours post challenge drug administration
  On the 4 dosing days, opioid withdrawal will be measured using the Clinical Opiate Withdrawal Scale (COWS) and the Subjective Opioid Withdrawal Scale (SOWS) at the following time points: 30 minutes pre-medication, 150 minutes post medication, 15 minutes post-challenge drug administration, 1 hour post- challenge drug administration, 2 hours post challenge drug administration and 3.5 hours post challenge drug administration

SECONDARY OUTCOMES:
Opioid Intoxication | 30 minutes pre-medication, 150 minutes post medication, 15 minutes post-challenge drug administration, 1 hour post- challenge drug administration, 2 hours post challenge drug administration and 3.5 hours post challenge drug administration
  On the 4 dosing days, opioid intoxication will be measured using the Visual Anaglog Scale (VAS)at the following time points: 30 minutes pre-medication, 150 minutes post medication, 15 minutes post-challenge drug administration, 1 hour post- challenge drug administration, 2 hours post challenge drug administration and 3.5 hours post challenge drug administration
Neuro-economic Choice Procedure | 45 minutes post challenge drug dosing
  A neuro-economics collaborative team will perform a neuro-economic choice paradigm procedure at 45 minutes post challenge drug dosing to determine the relative proportion and amount of a further dose of drug at 3.5 hours post challenge drug administration versus receipt of a variable amount of money

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ross, MD, Principal Investigator — NYU School of Medicine & Bellevue Hospital Center
Locations (1):
- Bellevue Hospital Center & the NYU School of Medicine, New York, New York, United States